CLINICAL TRIAL: NCT00253396
Title: THE PRISM Study-Low-Molecular-Weight Heparin Versus Unfractionated Heparin for Perioperative Bridging Anticoagulation: the Patient Preference for Self-Injection Study and Related Measurements
Brief Title: Patients Preference With Self-Injection: The PRISM Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: St. Joseph's Health Care London (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-2482
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2007-05

CONDITIONS: Bruises
Keywords: warfarin; clinical trial; pain measurement; heparin; heparin, low-molecular-weight; Anticoagulants
MeSH Terms: conditions — Contusions | interventions — Heparin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Unfractionated heparin
Drug: Enoxaparin

SUMMARY:
The purpose of this study is to determine which short-acting blood thinner (low-molecular-weight heparin [Enoxaparin] or unfractionated heparin) is associated with less discomfort and bruising when given as a subcutaneous (under the skin) injection before and after a planned surgery or procedure in patients who temporarily stop warfarin.

DETAILED DESCRIPTION:
Increasing Patient Comfort and Compliance: The Bridging Anticoagulation Clinic strives to provide the highest quality of care to patients who require temporary interruption of warfarin therapy. An important component of optimizing patient care is minimizing patient discomfort with perioperative administration of short-acting anticoagulants (LWMH or UFH) used for bridging therapy, which, in turn, may optimize patient compliance with this treatment. This issue is especially relevant for patients who are receiving out-of-hospital treatment with LMWH or UFH because about 85% of such patients will be taught to self-administer this medication. This study seeks to determine if there is less discomfort and bruising associated with self-injection of LMWH than with UFH.

Minimizing Injection Site Bruising: No studies, to our knowledge, have assessed the characteristics or clinical importance of bruising in patients receiving subcutaneous LMWH or UFH. Thus, there is no evidence to support any association between bruising and discomfort. To bridge this gap in knowledge, we will document each injection site during the course of the study and measure the amount of bruising observed using a standardized photographic methodology. Injection site bruising has the potential to cause medical problems if an injection site hematoma develops, which can become infected or can cause long-term discomfort.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is receiving warfarin therapy with a target international normalized ratio (INR) of 2.0-3.5
2. Patient requires temporary interruption of warfarin because of elective surgery or procedure.

Exclusion Criteria:

1. History of allergy to heparin, including heparin-induced thrombocytopenia (HIT)
2. Bridging anticoagulation with low molecular weight heparin (LMWH) or unfractionated heparin (UFH) not indicated
3. Impaired cognitive function or language barrier
4. Creatinine clearance < 30 ml/min
5. Patient declines consent
6. Patient is < 18 years of age.
7. Patient is not willing and able to self inject.
8. Patient has significant visual or hand motor impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Study Completion 2007-01

PRIMARY OUTCOMES:
The primary outcome measure is self-reported comfort score based on a visual analogue scale (VAS). Patients will complete a 10-point VAS. Patients will complete a VAS at the time of injection.

SECONDARY OUTCOMES:
On the day of the procedure, bruising at injection sites will be evaluated.
Patients will document in a diary each injection before and after the surgery or invasive procedure. On the day of surgery or procedure abdominal bruising measurement will be obtained. A digital photo will be take of the injection site.

CONTACTS AND LOCATIONS:
Overall Officials: Co-Investigators Dr. James Douketis and Karen Woods RN, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Background] McConnell EA. Administering subcutaneous heparin. Nursing. 2000 Jun;30(6):17. doi: 10.1097/00152193-200030060-00004. No abstract available. PMID 10865654
- [Result] Letizia M, Shenk J, Jones TD. Intermittent subcutaneous injections of pain medication: effectiveness, manageability, and satisfaction. Am J Hosp Palliat Care. 1999 Jul-Aug;16(4):585-92. doi: 10.1177/104990919901600407. PMID 10661066
- [Result] Martin S, Jones JS, Wynn BN. Does warming local anesthetic reduce the pain of subcutaneous injection? Am J Emerg Med. 1996 Jan;14(1):10-2. doi: 10.1016/S0735-6757(96)90003-0. PMID 8630132
- [Result] Hadley SA, Chang M, Rogers K. Effect of syringe size on bruising following subcutaneous heparin injection. Am J Crit Care. 1996 Jul;5(4):271-6. PMID 8811149
- [Result] Douketis JD. Perioperative anticoagulation management in patients who are receiving oral anticoagulant therapy: a practical guide for clinicians. Thromb Res. 2002 Oct 1;108(1):3-13. doi: 10.1016/s0049-3848(02)00387-0. PMID 12586125
- [Result] Dunn AS, Turpie AG. Perioperative management of patients receiving oral anticoagulants: a systematic review. Arch Intern Med. 2003 Apr 28;163(8):901-8. doi: 10.1001/archinte.163.8.901. PMID 12719198
- [Result] Jaffer AK, Brotman DJ, Chukwumerije N. When patients on warfarin need surgery. Cleve Clin J Med. 2003 Nov;70(11):973-84. doi: 10.3949/ccjm.70.11.973. PMID 14650471
- [Result] Spyropoulos AC, Jenkins P, Bornikova L. A disease management protocol for outpatient perioperative bridge therapy with enoxaparin in patients requiring temporary interruption of long-term oral anticoagulation. Pharmacotherapy. 2004 May;24(5):649-58. doi: 10.1592/phco.24.6.649.34740. PMID 15162899
- [Result] Hirsh J, Warkentin TE, Shaughnessy SG, Anand SS, Halperin JL, Raschke R, Granger C, Ohman EM, Dalen JE. Heparin and low-molecular-weight heparin: mechanisms of action, pharmacokinetics, dosing, monitoring, efficacy, and safety. Chest. 2001 Jan;119(1 Suppl):64S-94S. doi: 10.1378/chest.119.1_suppl.64s. No abstract available. PMID 11157643
- [Result] Dolovich LR, Ginsberg JS, Douketis JD, Holbrook AM, Cheah G. A meta-analysis comparing low-molecular-weight heparins with unfractionated heparin in the treatment of venous thromboembolism: examining some unanswered questions regarding location of treatment, product type, and dosing frequency. Arch Intern Med. 2000 Jan 24;160(2):181-8. doi: 10.1001/archinte.160.2.181. PMID 10647756
- [Result] Buller HR, Agnelli G, Hull RD, Hyers TM, Prins MH, Raskob GE. Antithrombotic therapy for venous thromboembolic disease: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):401S-428S. doi: 10.1378/chest.126.3_suppl.401S. PMID 15383479